CLINICAL TRIAL: NCT02275117
Title: A Parallel Group, Double-Blind, Randomized, Placebo Controlled, Dose-Ranging Phase 2 Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of ALD403 Administered Intravenously in Patients With Chronic Migraine
Brief Title: A Multicenter Assessment of ALD403 in Chronic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALD403-CLIN-005
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Migraine Disorders
Keywords: Migraine Disorders; ALD403
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- ALD403 Dose Level 1 (Experimental): ALD403 Dose Level 1 (IV)
  Interventions: Biological: ALD403
- ALD403 Dose Level 2 (Experimental): ALD403 Dose Level 2 (IV)
  Interventions: Biological: ALD403
- ALD403 Dose Level 3 (Experimental): ALD403 Dose Level 3 (IV)
  Interventions: Biological: ALD403
- ALD403 Dose Level 4 (Experimental): ALD403 Dose Level 4 (IV)
  Interventions: Biological: ALD403
- Placebo (Placebo Comparator): Placebo (IV)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALD403
  Other Names: Eptinezumab-jjmr; Vyepti
  Arms: ALD403 Dose Level 1; ALD403 Dose Level 2; ALD403 Dose Level 3; ALD403 Dose Level 4
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess ALD403 in the prevention of migraine headache in chronic migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine at ≤ 35 years of age with history of chronic migraine ≥ 1 year
* During the 28 day screening period, must have ≥ 15 headache days of which ≥ 8 days were assessed as migraine days with at least 5 migraine attacks as recorded in the eDiary
* Headache eDiary was completed on at least 22 of the 28 days prior to randomization

Exclusion Criteria:

* Confounding pain syndromes (e.g. fibromyalgia, chronic low back pain, complex regional pain syndrome) or any pain syndrome that requires regular analgesia
* Psychiatric conditions that are uncontrolled and untreated, including conditions that are not controlled for a minimum of 6 months prior to screening.
* History or diagnosis of complicated migraine (ICHD-III beta version, 2013), chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, migraine with brainstem aura, sporadic and familial hemiplegic migraine
* Unable to differentiate migraine from other headaches
* Subject has received botulinum toxin for migraine or for any other medical/cosmetic reasons requiring injections in the head, face, or neck within 4 months prior to screening.
* Have any clinically significant concurrent medical condition
* Receipt of any monoclonal antibody treatment within 6 months of screening (within or outside a clinical trial)
* Previously dosed with ALD403 or any monoclonal antibody targeting the CGRP pathway

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 665 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff TL Smith, MD, Study Director — Alder Biopharmaceuticals, Inc.
Locations (85):
- United States (78):
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Encino, California
  - Reserach Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Oakland, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Stanford, California
  - Research Site, Ventura, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evansville, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Brockton, Massachusetts
  - Research Site, New Bedford, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Princeton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Amherst, New York
  - Research Site, Brooklyn, New York
  - Research Site, Endwell, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Cary, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Orem, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Australia (3):
  - Research Site, Sydney, New South Wales
  - Research Site, Melbourne, Victoria
  - Research Site, Perth, Western Australia
- Research Site, Tbilisi, Georgia
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Hamilton

REFERENCES:
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Ettrup A, Shen V. Cardiovascular outcomes in adults with migraine treated with eptinezumab for migraine prevention: pooled data from four randomized, double-blind, placebo-controlled studies. J Headache Pain. 2021 Nov 25;22(1):143. doi: 10.1186/s10194-021-01360-1. PMID 34823467
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Schaeffler B, Shen V, Sperling B, Brevig T, Josiassen MK, Brunner E, Honeywell L, Mehta L. Safety and tolerability of eptinezumab in patients with migraine: a pooled analysis of 5 clinical trials. J Headache Pain. 2021 Mar 30;22(1):16. doi: 10.1186/s10194-021-01227-5. PMID 33781209
- [Derived] Dodick DW, Lipton RB, Silberstein S, Goadsby PJ, Biondi D, Hirman J, Cady R, Smith J. Eptinezumab for prevention of chronic migraine: A randomized phase 2b clinical trial. Cephalalgia. 2019 Aug;39(9):1075-1085. doi: 10.1177/0333102419858355. Epub 2019 Jun 24. PMID 31234642
- See also: Related Info — http://www.migrainestudynow.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1552 participants signed the ICF, of which 665 participants met the entry criteria and were randomized into the trial.
Groups:
- 300 mg ALD403: Participants were randomized to receive a single 300 mg IV infusion of ALD403 on Day 0
- 100 mg ALD403: Participants were randomized to receive a single 100 mg IV infusion of ALD403 on Day 0
- 30 mg ALD403: Participants were randomized to receive a single 30 mg IV infusion of ALD403 on Day 0
- 10 mg ALD403: Participants were randomized to receive a single 10 mg IV infusion of ALD403 on Day 0
- Placebo: Participants were randomized to receive a single placebo IV infusion on Day 0
Period: Overall Study
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Started | 131 | 133 | 134 | 133 | 134
Randomized and Treated (3 participants received duplicate randomization, participants are summarized in first group assigned) | 120 | 123 | 122 | 130 | 121
Completed | 97 | 96 | 92 | 100 | 98
Not Completed | 34 | 37 | 42 | 33 | 36
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 6 | 7 | 5 | 2 | 10
Not completed — Lost to Follow-up | 11 | 16 | 15 | 16 | 8
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 7 | 3 | 3
Not completed — Terminated by Sponsor | 4 | 4 | 4 | 6 | 4
Not completed — Worsening of Study Indication | 0 | 1 | 2 | 0 | 0
Not completed — Study Burden | 5 | 4 | 7 | 5 | 7
Not completed — Other | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population includes all subjects who received investigational product or placebo. 3 participants received duplicate randomization, participants are summarized within treatment group for which they actually received treatment.
Groups:
- 300 mg ALD403: Participants received a single 300 mg IV infusion of ALD403 on Day 0
- 100 mg ALD403: Participants received a single 100 mg IV infusion of ALD403 on Day 0
- 30 mg ALD403: Participants received a single 30 mg IV infusion of ALD403 on Day 0
- 10 mg ALD403: Participants received a single 10 mg IV infusion of ALD403 on Day 0
- Placebo: Participants received a single placebo IV infusion on Day 0
- Total: Total of all reporting groups
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo | Total
Number analyzed (Participants) | 121 | 122 | 122 | 130 | 121 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (10.0) | 36.7 (9.4) | 35.7 (9.4) | 36.4 (10.3) | 37.2 (9.2) | 36.6 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 104 | 111 | 113 | 109 | 535
  Male | 23 | 18 | 11 | 17 | 12 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 23 | 17 | 27 | 16 | 101
  Not Hispanic or Latino | 103 | 99 | 105 | 103 | 105 | 515
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 2 | 1 | 4
  Asian | 1 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 4 | 12 | 14 | 12 | 7 | 49
  White | 114 | 108 | 103 | 113 | 109 | 547
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 3 | 2 | 3 | 12
Region of Enrollment [Number; unit: participants]
  New Zealand | 7 | 1 | 0 | 1 | 2 | 11
  United States | 101 | 106 | 107 | 115 | 99 | 528
  Georgia | 11 | 9 | 14 | 9 | 15 | 58
  Australia | 2 | 6 | 1 | 5 | 5 | 19
Baseline Migraine Days [Count of Participants; unit: Participants] — Number of migraine days per month
  Participants
    < 20 days | 84 | 85 | 87 | 90 | 84 | 430
    ≥ 20 days | 37 | 37 | 35 | 40 | 37 | 186
Medication Overuse Status [Count of Participants; unit: Participants] — Investigator judgement of medication overuse status.
  Participants
    No | 56 | 62 | 57 | 64 | 57 | 296
    Yes | 65 | 60 | 65 | 66 | 64 | 320

OUTCOME MEASURES:

1. Primary Outcome: 75% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 75% over Weeks 1 to 12, as compared with baseline.
Time Frame: 12 Weeks
Population: Modified Full Analysis Population - Randomized participants who received investigational product or placebo, excluding participants from a site that was terminated by the Sponsor.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Participants | 38 | 37 | 33 | 33 | 24
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority — 75% Migraine Responder Rate - Week 1-12 (Modified Full Analysis Population); p = 0.0330, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.6, 95% CI 2-sided [1.3 to 24.0]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority — 75% Migraine Responder Rate - Week 1-12 (Modified Full Analysis Population); p = 0.0715, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [-0.5 to 21.8]
Statistical Analysis 3: Comparison: 30 mg ALD403 vs Placebo; Test type: Superiority — 75% Migraine Responder Rate - Week 1-12 (Modified Full Analysis Population); p = 0.2013, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [-3.5 to 18.5]
Statistical Analysis 4: Comparison: 10 mg ALD403 vs Placebo; Test type: Superiority — 75% Migraine Responder Rate - Week 1-12 (Modified Full Analysis Population); p = 0.2938, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 6.1, 95% CI 2-sided [-4.6 to 16.9]

2. Secondary Outcome: 50% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 50% over Weeks 1 to 12, as compared with baseline
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Participants | 65 | 65 | 65 | 54 | 47

3. Secondary Outcome: 50% Headache Responder Rate
Description: Participants with an average reduction in headache days of at least 50% over Weeks 1 to 12, as compared with baseline
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Participants | 59 | 55 | 55 | 48 | 39

4. Secondary Outcome: 100% Headache Responder Rate
Description: Participants with an average reduction in headache days of at least 100% over Weeks 1 to 12, as compared with baseline
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Participants | 4 | 0 | 0 | 1 | 1

5. Secondary Outcome: 100% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 100% over Weeks 1 to 12, as compared with baseline
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Participants | 9 | 6 | 5 | 10 | 3

6. Secondary Outcome: The Change From Baseline in Monthly Headache Days, Weeks 1-12
Description: Monthly headache days, as measured by eDiary. 4-weekly intervals averaged across weeks 1-12.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
days | -9.6 (6.94) | -8.9 (6.79) | -9.2 (6.33) | -7.5 (6.93) | -6.9 (6.37)

7. Secondary Outcome: The Change From Baseline in Monthly Migraine Days, Weeks 1-12
Description: Monthly migraine days, as measured by eDiary. 4-weekly intervals averaged across weeks 1-12.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
days | -8.2 (7.00) | -7.7 (6.87) | -7.9 (6.38) | -6.7 (6.80) | -5.6 (6.56)

8. Secondary Outcome: Change From Baseline in Percentage of Severe Migraines
Description: The change from baseline in percentage of migraines that are classified as severe over Weeks 1-12
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of severe migraines
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of severe migraines | -20.7 (29.47) | -15.9 (27.38) | -17.2 (26.98) | -16.1 (29.80) | -9.7 (27.32)

9. Secondary Outcome: Change From Baseline in Percentage of Severe Headaches
Description: The change from baseline in percentage of headaches that are classified as severe over Weeks 9-12
Time Frame: Weeks 9-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of severe headaches
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of severe headaches | -19.91 (25.800) | -10.36 (28.004) | -12.17 (30.197) | -11.42 (30.517) | -6.48 (27.211)

10. Secondary Outcome: The Change From Baseline to Week 12 in HIT-6 Total Score
Description: The HIT-6 measures the impact of headache on the participant's functional health and well-being in 6 domains: pain; role functioning (ability to carry out usual activities); social functioning; energy or fatigue; cognition; and emotional distress assessed over the prior 12-week period. The total possible scores range from 36 (no impact) to 78 (worst impact). A score of 60 or above is labeled as "severe".
Time Frame: Baseline to 12
Population: as for outcome 1
Measure: Number; unit: percentage of HIT-6 total score
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of HIT-6 total score | -60.4 | -43.4 | -34.9 | -34.8 | -28.4

11. Secondary Outcome: Percent Change From Baseline in Headache Days
Description: Monthly headache days, as measured by eDiary. 4-weekly intervals averaged across weeks 1-12.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of headache days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of headache days | -46.12 (31.481) | -43.09 (33.912) | -44.37 (28.620) | -37.20 (34.112) | -34.02 (30.970)

12. Secondary Outcome: Percent Change From Baseline in Migraine Days
Description: Monthly migraine days, as measured by eDiary. 4-weekly intervals averaged across weeks 1-12.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of migraine days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of migraine days | -48.88 (41.243) | -46.79 (40.983) | -46.74 (36.588) | -40.80 (40.133) | -35.37 (41.100)

13. Secondary Outcome: Time to First Migraine After Dosing
Description: The median number of days after dosing a participant had the next migraine using the eDiary as the recall method
Time Frame: Baseline to Week 49 (End of Study)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Days | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 5.0] | 3.0 [2.0 to 5.0] | 4.0 [3.0 to 5.0] | 2.0 [1.0 to 3.0]

14. Secondary Outcome: Change From Baseline in Monthly Migraine Attacks, Weeks 1-12
Description: The number of monthly migraine attacks summarized over Weeks 1-12. A migraine attack is defined as 1 continuously recorded migraine. One attack may result in multiple migraine days
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Migraine Attacks
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Migraine Attacks | -6.8 (5.4) | -6.5 (4.9) | -6.9 (5.0) | -6.2 (5.2) | -5.5 (5.0)

15. Secondary Outcome: Change From Baseline in Monthly Headache Episodes, Weeks 1-12
Description: The number of monthly headache episodes as summarized over Weeks 1-12. A headache episode is defined as 1 continuously recorded headache. One episode may result in multiple headache days
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Headache Episodes
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Headache Episodes | -8.2 (5.54) | -8.0 (5.37) | -8.3 (5.55) | -7.3 (5.37) | -7.0 (5.13)

16. Secondary Outcome: Change From Baseline in Monthly Migraine Hours, Weeks 1-12
Description: Migraine hours are the sum of the duration of migraines within 4 week intervals, and the average 4 week duration within 12 week intervals.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Migraine Hours
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Migraine Hours | -70.9 (100.34) | -64.2 (114.58) | -63.1 (84.56) | -49.2 (103.83) | -34.9 (100.87)

17. Secondary Outcome: Change From Baseline in Monthly Headache Hours, Weeks 1-12
Description: Headache hours are the sum of the duration of headaches within 4 week intervals, and the average 4 week duration within 12 week intervals.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Headache Hours
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
Headache Hours | -73.9 (101.53) | -60.9 (114.77) | -62.9 (81.89) | -47.5 (102.84) | -38.7 (99.26)

18. Secondary Outcome: Change From Baseline to Weeks 9-12 in Percentage of Migraines With Use of Acute Medication
Description: The percent of migraines with acute medication usage. Participants with no migraines will be included with a rate of zero.
Time Frame: Weeks 9-12
Measure: Mean (Standard Deviation); unit: percentage of acute medication migraines
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of acute medication migraines | -15.43 (39.121) | -10.36 (43.890) | -4.44 (37.746) | -10.03 (40.460) | -9.60 (37.451)

19. Secondary Outcome: Change From Baseline to Weeks 9-12 in Percentage of Headaches With Use of Acute Medication
Description: The percent of headaches with acute medication usage. Participants with no headaches will be included with a rate of zero.
Time Frame: Weeks 9-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of acute medication headaches
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
percentage of acute medication headaches | -5.98 (34.144) | -3.27 (34.419) | 1.52 (30.013) | -3.14 (32.853) | -3.42 (32.890)

20. Secondary Outcome: Baseline and Change From Baseline in Short Form Health Survey (SF-36, Version 2.0) at Week 12
Description: The SF-36 is a health survey containing 36 questions consisting of eight scaled scores to measure quality of life over the past 4 weeks (range: 0=worst to 100=best). Increases from baseline indicate improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SF-36 Score
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
Number analyzed (Participants) | 114 | 118 | 117 | 123 | 116
SF-36 Score
  Physical Functioning - Baseline | 50.5 (8.7) | 50.6 (7.8) | 51.1 (7.6) | 50.3 (8.4) | 50.2 (6.5)
  Physical Functioning - Week 12 | 53.6 (5.0) | 51.2 (8.3) | 52.5 (7.2) | 51.3 (7.9) | 51.9 (6.1)
  Role Physical - Baseline | 43.9 (9.5) | 45.2 (9.3) | 45.6 (9.3) | 44.9 (9.9) | 44.3 (9.6)
  Role Physical - Week 12 | 50.9 (7.2) | 48.9 (9.3) | 49.9 (7.7) | 47.9 (9.9) | 48.5 (8.3)
  Bodily Pain -Baseline | 42.7 (9.5) | 42.7 (9.6) | 44.5 (9.9) | 43.0 (9.6) | 42.5 (9.4)
  Bodily Pain - Week 12 | 48.9 (8.4) | 46.5 (9.9) | 48.1 (9.2) | 46.6 (9.3) | 46.0 (9.5)
  General Health - Baseline | 50.4 (9.2) | 50.7 (9.8) | 50.9 (8.7) | 51.1 (9.5) | 50.7 (9.8)
  General Health - Week 12 | 51.8 (8.7) | 50.7 (10.2) | 50.7 (9.2) | 52.7 (9.8) | 50.6 (10.0)
  Vitality - Baseline | 48.3 (8.9) | 50.1 (10.6) | 49.6 (9.8) | 49.4 (10.1) | 48.1 (10.9)
  Vitality - Week 12 | 51.3 (7.8) | 50.9 (10.5) | 50.6 (11.3) | 50.7 (10.6) | 51.1 (10.2)
  Social Functioning - Baseline | 45.0 (10.8) | 46.3 (10.1) | 46.8 (10.7) | 45.5 (10.4) | 45.4 (10.3)
  Social Functioning - Week 12 | 50.5 (8.1) | 48.7 (10.1) | 49.5 (9.0) | 47.7 (9.8) | 48.1 (8.7)
  Role Emotional - Baseline | 50.2 (9.1) | 49.4 (9.6) | 49.4 (9.7) | 49.8 (10.3) | 50.9 (8.1)
  Role Emotional - Week 12 | 51.4 (8.2) | 50.2 (9.0) | 51.2 (7.2) | 50.9 (8.4) | 51.0 (8.3)
  Mental Health - Baseline | 51.4 (8.4) | 52.0 (9.3) | 51.8 (9.5) | 51.4 (9.5) | 50.8 (9.8)
  Mental Health - Week 12 | 52.1 (8.8) | 50.8 (10.1) | 51.2 (9.5) | 52.2 (9.5) | 52.4 (8.8)
  Mental Component Score - Baseline | 50.4 (9.4) | 50.9 (9.7) | 50.5 (9.6) | 50.4 (9.9) | 50.5 (9.0)
  Mental Component Score - Week 12 | 51.2 (9.0) | 50.5 (9.7) | 50.7 (9.4) | 51.3 (9.3) | 51.5 (8.9)
  Physical Component Score - Baseline | 45.5 (8.4) | 46.1 (8.4) | 47.1 (7.7) | 46.1 (8.3) | 45.5 (7.9)
  Physical Component Score - Week 12 | 51.2 (6.8) | 49.0 (8.6) | 50.1 (7.0) | 48.8 (8.5) | 48.4 (8.1)

ADVERSE EVENTS:
Time Frame: Baseline to Week 49 (end of study)
Description: 3 participants received duplicate randomization, participants are summarized within treatment group for which they actually received treatment.
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | 30 mg ALD403 | 10 mg ALD403 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/122 | 0/122 | 0/130 | 0/121
Serious Adverse Events (participants affected / at risk) | 7/121 | 4/122 | 0/122 | 1/130 | 1/121
Other Adverse Events (participants affected / at risk) | 40/121 | 38/122 | 26/122 | 35/130 | 37/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=121) | 100 mg ALD403 (N=122) | 30 mg ALD403 (N=122) | 10 mg ALD403 (N=130) | Placebo (N=121)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vaginal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Serotonin syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Substance-induced mood disorders (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Menorrhagia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Pelvic pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Respiratory distress (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=121) | 100 mg ALD403 (N=122) | 30 mg ALD403 (N=122) | 10 mg ALD403 (N=130) | Placebo (N=122)
Nausea (Gastrointestinal disorders) | 8 | 9 | 4 | 6 | 9
Bronchitis (Infections and infestations) | 4 | 4 | 4 | 4 | 9
Nasopharyngitis (Infections and infestations) | 9 | 8 | 3 | 6 | 6
Sinusitis (Infections and infestations) | 8 | 3 | 6 | 8 | 6
Upper respiratory tract infection (Infections and infestations) | 13 | 8 | 7 | 9 | 6
Urinary tract infection (Infections and infestations) | 6 | 3 | 1 | 4 | 5
Dizziness (Nervous system disorders) | 2 | 12 | 3 | 11 | 9
Migraine (Nervous system disorders) | 1 | 7 | 3 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No